CLINICAL TRIAL: NCT02612051
Title: A FTIH Study With GSK3008348 in Healthy Volunteers and Patients With Idiopathic Pulmonary Fibrosis
Brief Title: First Time in Human (FTIH) Study of GSK3008348 in Healthy Volunteers and Idiopathic Pulmonary Fibrosis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200262
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: patients; FTIH; healthy volunteers; GSK3008348; [18F]-FBA-A20FMDV2; Idiopathic Pulmonary Fibrosis; PET
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part A, Cohort 1: GSK3008348 1-3000 mcg/Placebo (Experimental): Healthy subjects will receive single 3 ascending doses of GSK3008348 (ranging from 1 to 3000 microgram [mcg]) and matching placebo by nebulisation in one of the four treatment period according to randomization. There will be washout period of at least 6 days between the doses. Actual doses may involve either an increase or a decrease in the planned dose as well as a repeat of the previous.
  Interventions: Drug: GSK3008348 Nebuliser solution; Drug: Placebo Nebuliser solution
- Part A, Cohort 2: GSK3008348 1-3000 mcg/Placebo (Experimental): Healthy subjects will receive single 3 ascending doses of GSK3008348 (ranging from 1 to 3000 microgram [mcg]) and matching placebo by nebulisation in one of the four treatment period according to randomization. There will be washout period of at least 6 days between the doses. Actual doses may involve either an increase or a decrease in the planned dose as well as a repeat of the previous.
  Interventions: Drug: GSK3008348 Nebuliser solution; Drug: Placebo Nebuliser solution
- Part A, Cohort 3: GSK3008348 1-3000 mcg/Placebo (Experimental): Healthy subjects will receive single 3 ascending doses of GSK3008348 (ranging from 1 to 3000 microgram [mcg]) and matching placebo by nebulisation in one of the four treatment period according to randomization. There will be washout period of at least 6 days between the doses. Actual doses may involve either an increase or a decrease in the planned dose as well as a repeat of the previous.
  Interventions: Drug: GSK3008348 Nebuliser solution; Drug: Placebo Nebuliser solution
- Part B, Cohort 4: GSK3008348/Placebo, IPF, Period 2 PET Scan (Experimental): IPF subject will receive single dose of GSK3008348 (safe and tolerated dose as per cohort 1 to 3) or Placebo in two treatment periods according to randomization. There will be washout period of 6 to 28 days between the doses. Subjects will receive up to three microdose administrations of [18F]-FBA-A20FMDV2 for the PET scanning in period 2.
  Interventions: Drug: GSK3008348 Nebuliser solution; Drug: Placebo Nebuliser solution; Radiation: GSK26346763: ([18F]-FBA-A20FMDV2) IV infusion
- Part B, Cohort 5: GSK3008348/Placebo, IPF, Period 2 PET Scan (Experimental): IPF subject will receive single dose of GSK3008348 (safe and tolerated dose as per cohort 1 to 3) or Placebo in two treatment periods according to randomization. There will be washout period of 6 to 28 days between the doses. Subjects will receive up to three microdose administrations of [18F]-FBA-A20FMDV2 for the PET scanning in period 2.
  Interventions: Drug: GSK3008348 Nebuliser solution; Drug: Placebo Nebuliser solution; Radiation: GSK26346763: ([18F]-FBA-A20FMDV2) IV infusion
- Part B, Cohort 6: GSK3008348/Placebo, IPF, Period 2 PET Scan (Experimental): IPF subject will receive single dose of GSK3008348 (safe and tolerated dose as per cohort 1 to 3) or Placebo in two treatment periods according to randomization. There will be washout period of 6 to 28 days between the doses. Subjects will receive up to three microdose administrations of [18F]-FBA-A20FMDV2 for the PET scanning in period 2.
  Interventions: Drug: GSK3008348 Nebuliser solution; Drug: Placebo Nebuliser solution; Radiation: GSK26346763: ([18F]-FBA-A20FMDV2) IV infusion
- Part B, Cohort 7: GSK3008348/Placebo, IPF, Period 2 PET Scan (Experimental): IPF subject will receive single dose of GSK3008348 (safe and tolerated dose as per cohort 1 to 3) or Placebo in two treatment periods according to randomization. There will be washout period of 6 to 28 days between the doses. Subjects will receive up to three microdose administrations of [18F]-FBA-A20FMDV2 for the PET scanning in period 2.
  Interventions: Drug: GSK3008348 Nebuliser solution; Drug: Placebo Nebuliser solution; Radiation: GSK26346763: ([18F]-FBA-A20FMDV2) IV infusion
- Part C, Cohort 8: GSK3008348, IPF, PET Scan (Experimental): IPF subject will receive single dose of GSK3008348 (safe and tolerated dose as per Part B) in two treatment periods. There will be washout period of 6 to 14 days between the doses. Subjects will receive up to three microdose administrations of [18F]-FBA-A20FMDV2 for the PET scanning in both periods.
  Interventions: Drug: GSK3008348 Nebuliser solution; Radiation: GSK26346763: ([18F]-FBA-A20FMDV2) IV infusion

INTERVENTIONS:
Drug: GSK3008348 Nebuliser solution — Nebuliser solution formulated at 5000 mcg/mL with 5% mannitol, citric acid, sodium citrate and water for injection, pH adjusted using Hydrochloric acid or Sodium hydroxide to the target pH 5.4 +/- 0.4. 4 ml of diluted dose of appropriate concentration will be administered by nebulisation.
Drug: Placebo Nebuliser solution — 5% mannitol nebuliser solution. 4 ml of solution will be administered by nebulisation
  Arms: Part A, Cohort 1: GSK3008348 1-3000 mcg/Placebo; Part A, Cohort 2: GSK3008348 1-3000 mcg/Placebo; Part A, Cohort 3: GSK3008348 1-3000 mcg/Placebo; Part B, Cohort 4: GSK3008348/Placebo, IPF, Period 2 PET Scan; Part B, Cohort 5: GSK3008348/Placebo, IPF, Period 2 PET Scan; Part B, Cohort 6: GSK3008348/Placebo, IPF, Period 2 PET Scan; Part B, Cohort 7: GSK3008348/Placebo, IPF, Period 2 PET Scan
Radiation: GSK26346763: ([18F]-FBA-A20FMDV2) IV infusion — Formulated in 0.9% saline. The maximum amount of radioactivity injected during each PET scan will be 150 Megabecquerel (MBq) and maximum mass of [18F]-FBA-A20FMDV2 administered across all three administrations will be 100 mcg. Intravenous bolus infusion of 20 ml will be administered over about 30 seconds.
  Arms: Part B, Cohort 4: GSK3008348/Placebo, IPF, Period 2 PET Scan; Part B, Cohort 5: GSK3008348/Placebo, IPF, Period 2 PET Scan; Part B, Cohort 6: GSK3008348/Placebo, IPF, Period 2 PET Scan; Part B, Cohort 7: GSK3008348/Placebo, IPF, Period 2 PET Scan; Part C, Cohort 8: GSK3008348, IPF, PET Scan

SUMMARY:
GSK3008348 is an investigational drug, being developed by GlaxoSmithKline Research and Development Limited (the Sponsor, a pharmaceutical company based in the UK) for the treatment of Idiopathic Pulmonary Fibrosis (IPF). IPF is a rare and poorly understood disease that causes scarring of the lungs. The main symptoms are shortness of breath and a dry cough. Symptoms generally worsen over time and in some subjects may prove fatal. The cause of IPF is unknown.

This is a First Time in Human, Phase 1, 3-part study which is being carried out on behalf of the Sponsor by Quintiles. The primary purpose of Part A is to examine the safety and tolerability of single nebulised (a medicated spray) doses of GSK3008348 following inhalation in healthy volunteers. The secondary objective is to determine how and at what rate the body absorbs, distributes, breaksdown and eliminates the drug.

Parts B and C of this study will be in-patients with Idiopathic Pulmonary Fibrosis (IPF). The purpose of Part B and C is to examine the safety and tolerability, and how much of the drug binds to its target, following single nebulised (a medicated spray) doses of GSK3008348 following inhalation in patients with Idiopathic Pulmonary Fibrosis (IPF). The secondary objective is to determine how and at what rate the bodies of these patients absorbs, distributes, breaksdown and eliminates the drug.

The total duration of Part A will be 65 - 87 days, Part B 62 days and Part C 43 days.

ELIGIBILITY:
Inclusion Criteria:

Part A:

- Male and female subjects >= 18 years at the time of signing the consent form.

Parts B and C :

- Male subjects >= 45 years and female subjects >= 55 years at the time of signing the consent form.

Part A:

* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, 12-lead ECG and pulmonary function tests.
* A subject with a potentially clinically significant abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with FEV1, FVC and DLCO values outside the normal range may be included only if the investigator in consultation with the Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.

Parts B and C:

* Subject is ambulant and capable of attending a PET scan visit as an outpatient.
* Subjects will have a diagnosis of IPF as determined by a responsible and experienced chest physician and based on established criteria defined by the American Thoracic Society/European Respiratory Society Internationale Multidisciplinary Consensus Classification of the Idiopathic Interstitial Pnuemonias.
* FVC > 50 % predicted and DLCO > 50% predicted. Following a review of the safety data at the interim, these criteria may be altered to FVC > 50% predicted and DLCO > 40% predicted.

Part A:

- Body weight >=50 Kilogram (kg) and BMI within the range 19.0 - 35.0 kg/meter square (m^2) (inclusive).

Parts B and C:

* Body weight >=45 kg and BMI within the range 18.0 - 35.0 kg/m^2 (inclusive)
* Female subjects are eligible to participate if they are of non-childbearing potential defined as premenopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 month of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-international unit (MIU)/millilitre (ml) and estradiol > 141 picomole (pmol)/litre (l) is confirmatory (as a precaution a pregnancy test is conducted prior to dosing, a positive test leads to exclusion).
* Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until 90 days after the last dose of study medication. a. Vasectomy with documentation of azoospermia b. Male condom plus partner use of one of the contraceptive options below: i. Contraceptive subdermal implant that meets the Standard Operating Procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label ii. Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label iii. Oral Contraceptive, either combined or progestogen alone iv. Injectable progestogen v. Contraceptive vaginal ring vi. Percutaneous contraceptive patches This is an all-inclusive list of those methods that meet the following GlaxoSmithKline (GSK) definition of highly effective: having a failure rate of less than 1% per year when used consistently and correctly and, when applicable, in accordance with the product label. For non-product methods (e.g., male sterility), the investigator determines what is consistent and correct use. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in protocol

Exclusion Criteria:

* Alanine transaminase and bilirubin >1.5x5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or history of photosensitivity.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QT interval corrected for heart rate (QTc )> 450 millisecond (msec) or QTc > 480 msec in subjects with Bundle Branch Block
* Current upper or lower respiratory tract infection on admission to the clinical unit.

Parts B and C:

* History or suffers from claustrophobia or subject feels unable to lie flat and still on their back for a period of up to 2 hours in the PET/ CT scanner (note, one rest period will be allowed during the scan if required).
* Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations or occupational exposure resulting in radiation exposure greater than 10 millisievert (mSv) over the past 3 years or greater than 10 mSv in a single year including the proposed study. Clinical exposure from which the subject receives a direct benefit is not included in these calculations.
* Subjects with current IPF exacerbation, upper or lower respiratory tract infection.
* Subjects with severe co-existent chronic obstructive pulmonary disease (COPD), for example FEV1 < 60% predicted.

All Parts:

* Use of prohibited medication
* Subjects who are currently taking Pirfenidone or Nintedanib or who have received Pirfenidone or Nintedanib within the 30 days prior to the first dosing day will be excluded from the study.
* Subjects prescribed long-term continuous home oxygen therapy (those whose use of oxygen is intermittent and for symptom relief only are not excluded)
* History of alcohol consumption regularly in excess of: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C Ribonucleic acid (RNA) polymerase chain reaction (PCR) test is obtained.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Parts B and C:

* Previous or current exposure to animals that may harbour foot and mouth disease virus (FMDV2).
* Previous long term (>= 3 months) residence in a country where FMDV2 is endemic (such as certain areas of Africa, Asia and South America)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

PRIMARY OUTCOMES:
Part A: Number of participants with adverse events (AE) as a measure of safety and tolerability | Up to Day 33
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AE will be collected from the start of study treatment until the final follow-up visit.
Part A: Temperature as a measure of safety and tolerability | Up to Day 33
Part A: Systolic and diastolic blood pressure as a measure of safety and tolerability | Up to Day 33
Part A: Pulse rate and respiratory rate as a measure of safety and tolerability | Up to Day 33
Part A: Peripheral capillary oxygen saturation (SpO2) levels as a measure of safety and tolerability | Up to Day 33
  SpO2 levels are estimates of the amount of oxygen in the blood. SpO2 will be measured by pulse oximetry.
Part A: ECG and Telemetry as a measure of safety and tolerability | Up to Day 21
  12-lead ECG and cardiac telemetry will be performed.
Part A: FEV1 and FVC as a measure of safety and tolerability | Up to Day 33
  Forced expiratory volume in 1 second (FEV1) is the volume of air that can forcibly be blown out in one second, after full inspiration. Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration. Lung function test will be performed to obtain FEV1 and FVC .
Part A: DLCO as a measure of safety and tolerability | Up to Day 20
  Diffusing capacity (DLCO) is the carbon monoxide uptake from a single inspiration in a standard time (usually 10 seconds). Lung function test will be performed to obtain DLCO.
Part A: Taste questionnaire for taste of nebulised GSK3008348 as a measure of safety and tolerability | Up to Day 19
  Subjects will be required to complete a taste questionnaire following dosing.
Part A: Composite of hematology laboratory tests as a measure of safety and tolerability | Up to Day 33
  Hematology laboratory tests will include platelet count, red blood cell count, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, neutrophils, lymphocytes, monocytes, eosinophils and basophils.
Part A: Composite of clinical chemistry laboratory tests as a measure of safety and tolerability | Up to Day 33
  Clinical chemistry laboratory tests will include urea, creatinine, glucose non-fasted, creatinine phosphokinase, potassium, sodium, calcium, aspartate aminotransferase alanine transaminase,total and direct bilirubin, total protein, alkaline phosphatise and albumin.
Part A: Composite of urinalysis laboratory tests as a measure of safety and tolerability | Up to Day 33
  Urinalysis laboratory tests will include specific gravity, pH, glucose, protein, blood and ketones by dipstick, microscopic examination (if blood or protein is abnormal).
Part B: AE as a measure of safety and tolerability | Up to Day 43
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AE will be collected from the start of study treatment until the final follow-up visit.
Part B: Temperature as a measure of safety and tolerability | Up to Day 43
Part B: Systolic and diastolic blood pressure as a measure of safety and tolerability | Up to Day 43
Part B: Pulse rate and respiratory rate as a measure of safety and tolerability | Up to Day 43
Part B: SpO2 levels as a measure of safety and tolerability | Up to Day 43
  SpO2 levels are estimates of the amount of oxygen in the blood. SpO2 will be measured by pulse oximetry.
Part B: ECG and Telemetry as a measure of safety and tolerability | Up to Day 31
  12-lead ECG and cardiac telemetry will be performed.
Part B: FEV1 and FVC as a measure of safety and tolerability | Up to Day 43
  FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. FVC is the volume of air that can forcibly be blown out after full inspiration. Lung function test will be performed to obtain FEV1 and FVC .
Part B: DLCO as a measure of safety and tolerability | Up to Day 30
  DLCO is the carbon monoxide uptake from a single inspiration in a standard time (usually 10 seconds). Lung function test will be performed to obtain DLCO.
Part B: Taste questionnaire for taste of nebulised GSK3008348 as a measure of safety and tolerability | Up to Day 29
  Subjects will be required to complete a taste questionnaire following dosing.
Part B: Changes in volume of distribution [VT]) at approximately 1 hour post-dose compared to pre-dose of [18F]-FBA-A20FMDV2 in the lung | Baseline (from Day 15), Up to Day 30
  Positron Emission Tomography (PET) scan and a sample of blood will be taken simultaneously for measurement of [18F]-FBA-A20FMDV2 concentration. The blood volume in tissue will be determined by dividing the tissue tracer concentration by the blood value. Changes in the uptake of [18F]-FBA-A20FMDV2 in the lung will be calculated.
Part B: Composite of hematology laboratory tests as a measure of safety and tolerability | Up to Day 30
  Hematology laboratory tests will include platelet count, red blood cell count, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, neutrophils, lymphocytes, monocytes, eosinophils and basophils.
Part B: Composite of clinical chemistry laboratory tests as a measure of safety and tolerability | Up to Day 30
  Clinical chemistry laboratory tests will include urea, creatinine, glucose fasted, creatinine phosphokinase, potassium, sodium, calcium, aspartate aminotransferase alanine transaminase, total and direct bilirubin, total protein, alkaline phosphatise and albumin.
Part B: Composite of urinalysis laboratory tests as a measure of safety and tolerability | Up to Day 30
  Urinalysis laboratory tests will include specific gravity, pH, glucose, protein, blood and ketones by dipstick, microscopic examination (if blood or protein is abnormal)
Part C: Changes in VT at various time points post-dose compared to pre-dose of [18F]-FBA-A20FMDV2 in the lung | Baseline (from Day 1), Up to Day 29
  PET scan and a sample of blood will be taken simultaneously for measurement of [18F]-FBA-A20FMDV2 concentration. The blood volume in tissue will be determined by dividing the tissue tracer concentration by the blood value. Changes in the uptake of [18F]-FBA-A20FMDV2 in the lung will be calculated.

SECONDARY OUTCOMES:
Part A: Area under the curve (AUC) following single doses of GSK3008348 | Blood samples will be collected at pre-dose and at 5, 10, 15, 30 minutes (mins), 1, 2, 3, 4, 6, 8, 12 hours (Day 1) and 24 hours (Day 2) post-dose of each treatment period
  AUC from time zero to infinity (AUC[0-inf]), AUC from time zero to the time of last quantifiable concentration (AUC[0-t]) will be calculated from concentration-time curve using the linear trapezoidal rule based on each individual subject's profile.
Part A: Cmax following single doses of GSK3008348 | Blood samples will be collected at pre-dose and at 5, 10, 15, 30 mins, 1, 2, 3, 4, 6, 8, 12 hours (Day 1) and 24 hours (Day 2) post-dose of each treatment period
  Maximum observed concentration (Cmax) will be calculated from concentration-time curve based on each individual subject's profile.
Part A: Tmax and t½ following single doses of GSK3008348 | Blood samples will be collected at pre-dose and at 5, 10, 15, 30 mins, 1, 2, 3, 4, 6, 8, 12 hours (Day 1) and 24 hours (Day 2) post-dose of each treatment period
  Time of maximum concentration (tmax) will be calculated from concentration-time curve based on each individual subject's profile. Elimination half-life (t½) is time required for or drug in the body to reduced by one-half. t½ will be calculated from concentration-time curve based on each individual subject's profile.
Part B: Area under the curve (AUC) following single doses of GSK3008348 | Blood samples will be collected at pre-dose and at 5, 10, 15, 30 mins, 1, 2, 3, 4, 6, 8, 12 hours (Day 1) and 24 hours (Day 2) post-dose of each treatment period
  AUC from time zero to infinity (AUC[0-inf]), AUC from time zero to the time of last quantifiable concentration (AUC[0-t]) will be calculated from concentration-time curve using the linear trapezoidal rule based on each individual subject's profile.
Part B: Cmax following single doses of GSK3008348 | Blood samples will be collected at pre-dose and at 5, 10, 15, 30 mins, 1, 2, 3, 4, 6, 8, 12 hours (Day 1) and 24 hours (Day 2) post-dose of each treatment period
  Maximum observed concentration (Cmax) will be calculated from concentration-time curve based on each individual subject's profile.
Part B: Tmax and t½ following single doses of GSK3008348 | Blood samples will be collected at pre-dose and at 5, 10, 15, 30 mins, 1, 2, 3, 4, 6, 8, 12 hours (Day 1) and 24 hours (Day 2) post-dose of each treatment period
  Time of maximum concentration (tmax) will be calculated from concentration-time curve based on each individual subject's profile. Elimination half-life (t½) is time required for or drug in the body to reduced by one-half. t½ will be calculated from concentration-time curve based on each individual subject's profile.
Part B: Changes in VT at 14-28 hours post-dose compared to pre-dose of [18F]-FBA-A20FMDV2 in the lung | Baseline (from Day 15), Up to Day 30
  PET scan and a sample of blood will be taken simultaneously for measurement of [18F]-FBA-A20FMDV2 concentration. The blood volume in tissue will be determined by dividing the tissue tracer concentration by the blood value. Changes in the uptake of [18F]-FBA-A20FMDV2 in the lung will be calculated.
Part C: Area under the curve (AUC) following single doses of GSK3008348 | Blood samples will be collected at pre-dose and post-nebulisation at 5, 10, 15, 30 mins, 1, 2, 3, 4, 6, 8, 12 hours (Day 1) and 24 hours (Day 2) post-dose of each treatment period
  AUC from time zero to infinity (AUC[0-inf]), AUC from time zero to the time of last quantifiable concentration (AUC[0-t]) will be calculated from concentration-time curve using the linear trapezoidal rule based on each individual subject's profile.
Part C: Cmax following single doses of GSK3008348 | Blood samples will be collected at pre-dose and post-nebulisation at 5, 10, 15, 30 mins, 1, 2, 3, 4, 6, 8, 12 hours (Day 1) and 24 hours (Day 2) post-dose of each treatment period
  Maximum observed concentration (Cmax) will be calculated from concentration-time curve based on each individual subject's profile.
Part C: Tmax and t½ following single doses of GSK3008348 | Blood samples will be collected at pre-dose and post-nebulisation at 5, 10, 15, 30 mins, 1, 2, 3, 4, 6, 8, 12 hours (Day 1) and 24 hours (Day 2) post-dose of each treatment period
  Time of maximum concentration (tmax) will be calculated from concentration-time curve based on each individual subject's profile. Elimination half-life (t½) is time required for or drug in the body to reduced by one-half. t½ will be calculated from concentration-time curve based on each individual subject's profile.
Part C: AE as a measure of safety and tolerability | Up to Day 43
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AE will be collected from the start of study treatment until the final follow-up visit.
Part C: Temperature as a measure of safety and tolerability | Up to Day 43
Part C: Systolic and diastolic blood pressure as a measure of safety and tolerability | Up to Day 43
Part C: Pulse rate and respiratory rate as a measure of safety and tolerability | Up to Day 43
Part C: Peripheral capillary oxygen saturation (SpO2) levels as a measure of safety and tolerability | Up to Day 43
  SpO2 levels are estimates of the amount of oxygen in the blood. SpO2 will be measured by pulse oximetry.
Part C: Composite of hematology laboratory tests as a measure of safety and tolerability | Up to Day 43
  Hematology laboratory tests will include platelet count, red blood cell count, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, neutrophils, lymphocytes, monocytes, eosinophils and basophils.
Part C: Composite of clinical chemistry laboratory tests as a measure of safety and tolerability | Up to Day 43
  Clinical chemistry laboratory tests will include urea, creatinine, glucose fasted, creatinine phosphokinase, potassium, sodium, calcium, aspartate aminotransferase alanine transaminase,, total and direct bilirubin, , total protein, alkaline phosphatise and albumin.
Part C: Composite of urinalysis laboratory tests as a measure of safety and tolerability | Up to Day 43
  Urinalysis laboratory tests will include specific gravity, pH, glucose, protein, blood and ketones by dipstick, microscopic examination (if blood or protein is abnormal)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study 200262 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/200262?search=study&b'search_terms=200262'#rs